CLINICAL TRIAL: NCT04853888
Title: Attachment and Child Health (ATTACH™) Program: Promoting Vulnerable Children's Health at Scale
Brief Title: ATTACH™ Program: Promoting Vulnerable Children's Health at Scale
Acronym: ATTACH™
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Nicole Letourneau, Chair in Parent-Infant Mental Health. Professor, Faculty of Nursing & Cumming School of Medicine (Pediatrics, Psychiatry & Community Health Sciences), Director of RESOLVE Alberta, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB20-0903
Record Dates: First submitted 2021-03-22; First posted 2021-04-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Parent-Child Relations
Keywords: Parent Child Interaction Quality; Parental Reflective Function; Child Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Other): * A quasi-experimental design was selected to more closely approximate service delivery models in agencies that do not typically employ control groups.
  * Given promising findings (from seven ATTACH™ pilot studies), a randomized controlled trial design, even employing wait-list controls was deemed unacceptable and even unethical by patients, health care professionals and health system administrators in engagement activities surrounding the preparation of this proposal.
  Interventions: Behavioral: ATTACH™ Parenting Program

INTERVENTIONS:
Behavioral: ATTACH™ Parenting Program — ATTACH™ parenting program offers an innovative, novel approach to early intervention, focusing on improving parent-child relationship quality by targeting parents' underlying reflective function (RF)-the ability to better understand one's own and one's child's thoughts and feelings. RF is essential for high quality parent-child relationships and secure parent-child attachment, both tied to child development and health, especially cognition, communication and inflammation.
  .

SUMMARY:
ATTACH™ is a psycho-educational parenting program, designed with community agencies serving families of preschoolers affected by toxic stress (e.g. parental depression, addictions, domestic violence, poverty) to bolster children's health and development. It focuses on improving parent-child relationship quality by targeting parents' reflective function (RF), i.e. the ability to better understand one's own and one's child's thoughts and feelings. RF is essential for high quality parent-child relationships and secure attachment, both tied to child development and health, especially cognition, communication and inflammation. ATTACH™ was implemented and tested in seven rapid-cycling pilot studies by researchers, guided by the IDEAS (Innovate, Develop, Evaluate, Adapt, Scale) Framework™, an innovative clinical trial approach. ATTACH™ significantly improved: (a) parent-child relationship quality and attachment, (b) parents' RF scores, and (c) children's cognitive and motor development. However, whether ATTACH™ continues to work with delivery by trained agency healthcare professionals rather than study researchers, in naturalistic, community settings remains to be seen. Small sample sizes also limited the ability to assess longer-term impacts and whether ATTACH™ is equally effective across patient populations. Further, another parenting intervention successfully reduced systemic inflammation in children exposed to toxic stress. Whether ATTACH™ impacts novel biomarkers of inflammation (i.e. immune cell gene expression and DNA methylation) is not known.

DETAILED DESCRIPTION:
Methods: This study is comprised of a pre/ post-test quasi-experimental design evaluation of the ATTACH™ program as well as an examination of implementation feasibility via Normalization Process Theory (NPT). While Objective 1 will be addressed first, Objective 2 will begin soon after so that information gathered in Objective 2 may be used to tailor the implementation in Objective 1 as appropriate.

Research Question & Objectives: The proposed research has the following two (quantitative and qualitative) arms: Objective 1 (Quantitative component): To evaluate community agencies delivered ATTACH™ impacts on: (1a) parent-child relationship quality, parental RF and child development, (1b) different patient populations (for whom program works best/worst), (1c) immune biomarkers indicative of inflammatory disease risk, i.e. gene expression and DNA methylation, (1d) health professionals' adherence to ATTACH™ program, via fidelity assessment, and (1e) outcomes 3 months post-intervention. Objective 2 (Qualitative component): To evaluate health care professionals' and administrators' perceptions and experiences of: (2a) intervention uptake and fidelity, (2b) implementation benefits, facilitators, barriers and challenges, and (2c) utility of ATTACH™ e-learning platform. The study participants can not be enrolled in the program without being in the research.

Objective 1: A quasi-experimental design was selected to more closely approximate service delivery models in agencies that do not typically employ control groups. We will intervene with 100 new patients and their birth to 36 month-old children, a sufficient sample size to detect minimum effect size (d=.34) for pre-intervention/post-intervention differences from the primary outcome of parent-child relationship quality, from the five community agencies. We plan to recruit 20 families (including parents, co-parents and children) from each agency.

Objective 2: NPT is used to uncover factors that interfere with the routine incorporation of interventions into health care. Thus, NPT is the ideal theory to guide our approaches including qualitative semi-structured interviews and analyses. NPT will enable the exploration of patients', health care professionals' and health system administrators' perceptions and experiences of intervention uptake and fidelity as well as the benefits, facilitators, barriers and challenges to ATTACH™ implementation by community agencies, including perceptions of the fidelity assessment tool and e-learning training.

Setting: Settings include Alcove Addiction Recovery, CUPS Calgary, Discovery House Women's Shelter, Sonshine Community Centre, and Steinbach Family Resource Centre, MB. Other interested agencies will also be involved. Patients, health care professionals and administrators from each agency will be recruited via convenience sampling methods to take part in one-on-one interviews. We plan to recruit 20 patients, 20 health care professionals and 20 administrators (total n= 60) at the participating agencies. However recruitment and data collection will continue until theoretical data saturation, i.e. the degree to which new data repeats or is redundant with what was expressed in previous data. We will employ a stopping rule: Data collection in a category (patient, health care professional, and health care administrator) will cease when three interviews in a row offer less than 5% new information. Only deidentified data will be sent by the participating agencies. Basic demographic data will be collected from stakeholders (patients, health care professionals, and administrators), including age, sex, employment and education. Using NPT in implementing complex interventions like ATTACH™, requires development of an interview guide addressing the four NPT concepts: coherence (meaning and sense making of ATTACH™ by participants), cognitive participation (commitment and engagement by participants), collective action (work the participants do to make ATTACH™ function), and reflexive monitoring (reflection of ATTACH™).

In finalizing the interview guide and developing the interview processes (e.g. home or clinic setting, telephone/web-conference, Zoom or in-person), the Patient Engagement Committee (PEC) and Community Engagement Committee (CEC) members will be engaged in review, feedback and decision making. The interview guide will be used for staff and patients and will be pilot tested before use. Interviews will be audio-recorded and transcribed verbatim with appropriate privacy protections in place to guard participant identity and personal information. Data analysis will occur in two parts. First, interviews will be transcribed and coded as soon as interviews are completed and examined for "nuggets" or key learnings that offer guidance to implementation in agencies. These nuggets will be shared with the Executive Team, PEC and CEC (especially relevant agency health care professionals and administrators) and discussed so that appropriate adjustments may be made to facilitate ATTACH™ normalization in agencies. Second, all transcripts will be coded using the stages of thematic analysis including familiarization, coding, theme development and data reporting. Theme and sub-theme development will be deductive, using a priori codes dictated by interview questions in order to explain factors that promote or inhibit interventions from being embedded in agency practice. As new interviews are undertaken, data will be examined to determine degree of data saturation. Two trainees will code the data, supervised by Letourneau, who is experienced in qualitative data analysis. Inter-rater reliability will be assessed and reported with Cohen's kappa coefficients; disagreements will be resolved by consensus. Data will be managed with QSR International NVivo12. Once themes and sub-themes are finalized, findings will be summarized in a draft report and shared with key informants as a validation check.

ELIGIBILITY:
Inclusion Criteria:

* parents with children between birth and 32 months of age (based on selection of age-appropriate tools for assessing children's health and development)
* parents agree to participate in the ATTACH™ program consisting of 10-12 weeks of one-hour per week parent training sessions
* parents agreed to bring a co-parent for 2-3 of the 10 sessions (when possible)
* parents agree to the dried blood sample collection from themselves and their children (in Calgary agencies)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Parent-Child Relationship Quality will be measured by Parent Child Interaction Teaching Scale (PCITS). | Change from baseline PCITS scores after completion of intervention and at 3 months.
  The PCITS scale (Sumner & Spietz, 1994) is an observational binary measure of interactions in parent-child teaching situations to measure parent-child interaction quality in infants 36 months or younger. Considered as the gold standard, PCITS consists of 73 items categorized into 6 subscales including parental sensitivity to cues, responsiveness to distress, growth fostering, and cognitive growth fostering, and infant clarity of cues and responsiveness to parent. Certified coders code the items either as yes or no; Yes responses are then summed to yield a total score for each sub-scale. Final PCITS scores include total scores for each subscale, parent total, child total, and parent-child total scores, along with total parent contingency and child contingency scores. The observation of teaching interaction typically takes 5 minutes. Scale range from 0 - 73. A higher score means a better outcome, i.e. higher quality of parent-child interaction.

SECONDARY OUTCOMES:
Parental Reflective Function will be measured by Parental Reflective Function Questionnaire (PRFQ). | Change from baseline PRFQ scores after completion of intervention and at 3 months.
  The PRFQ (Luyten et al., 2017) is an 18-item self-reported questionnaire that assesses parental RF and takes 5 minutes to administer. It consists of 3 subscales to capture key features of parental RF including: (a) Pre-mentalizing subscale to assess non-mentalizing modes characteristic of parents with impairments in RF (b) Certainty in Mental States subscale to examine the capacity to recognize the opacity of mental states, and (c) Interest and Curiosity subscale that relates to parental interest and curiosity in mental states. Each subscale consists of 6 items and each item is rated on a 7-point Likert scale. For the PRFQ Pre-mentalizing subscale, higher scores indicate lower levels of parental RF . For the PRFQ Certainty in Mental States and Interest and Curiosity subscales, average levels of both PRFQ Certainty in Mental States and Interest and Curiosity subscales may be most adaptive, whereas either low or very high levels may be more maladaptive.
Child Development, measured by Ages and Stages Questionnaire - 3rd Edition | Change from baseline ASQ-3 scores after completion of intervention and at 3 months.
  Developed by Squires and Bricker (2009), ASQ - 3 is a series of parent-completed questionnaires to assess child development in 5 domains namely communication, gross motor, fine motor, problem solving, and personal-social skills. There are 21 versions for different age groups 21 ranging from 1 to 66 months, with 6 questions in each domain asking if the child can or cannot do age-appropriate tasks. Adding up items in each domain provides a total score for that domain (Mackrides, 2011). Summing up total scores for each domain yields the total score (out of 60). Higher scores are indicative of healthier outcomes (Bedford, 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Letourneau, PhD RN FCAHS, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anis L, Letourneau N, Ross KM, Hart M, Graham I, Lalonde S, Varro S, Baldwin A, Soulsby A, Majnemer A, Donnelly C, Piotrowski C, Collier C, Lindeman C, Goldowitz D, Isaac D, Thomson D, Serre D, Citro E, Zimmermann G, Pliszka H, Mann J, Baumann J, Piekarski J, Dalton JA, Johnson-Green J, Wood K, Bruce M, Santana M, Mayer M, Gould M, Kobor M, Flowers M, Haywood M, Koerner M, Parker N, Muhajarine N, Fairie P, Chrishti R, Perry R, Merrill S, Pociuk S, StephanieTaylor, Cole S, Murphy T, Marchment T, Xavier V, Shajani Z, West Z. Study protocol for Attachment & Child Health (ATTACHTM) program: promoting vulnerable Children's health at scale. BMC Pediatr. 2022 Aug 19;22(1):491. doi: 10.1186/s12887-022-03439-3. PMID 35986306